CLINICAL TRIAL: NCT02894437
Title: Qualitative Study of Preventive Organization of the Pelvic Bedsores Injured Spinal Cord: Building a Conceptual Framework Based on the Perceptions and Behaviors of Patients and Professionals Involved
Brief Title: Qualitative Study of Preventive Organization of the Pelvic Bedsores Injured Spinal Cord
Acronym: QUALIPREPS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0023
Record Dates: First submitted 2016-08-11; First posted 2016-09-09 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Spinal Cord Injuries; Pressure Ulcers
Keywords: prevention; organization; pressure ulcers
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients: SCI recruited Physical Medicine and Nantes University Hospital Rehabilitation. Recruitment will try to balance the number of people in four sub-groups followed and complicated (= history of pelvic pressure sores), not followed and uncomplicated, monitored and uncomplicated, not followed and complicated
  Interventions: Other: qualitative interviews
- health professionals: those involved in the chain of care Spinal Cord concerning various professions (including medical, paramedical and administrative) decision and variable influence on the organization of the die care of spinal injuries.
  Interventions: Other: qualitative interviews

INTERVENTIONS:
Other: qualitative interviews — semi-structured interviews as a conceptual frame work

SUMMARY:
The purpose of the Protocol is the prevention of pelvic pressure ulcers within a care network of SCI patients whose general organization refers to the medical literature and the recommendations of the ministerial circular of 18 June 2004. A conceptual framework for work (CFW) will be set up and semi-structured interviews will be conducted with patients and professionals. They will confirm or dismiss the CFW gradually with a refined coding As of domains and sub-domains of the skin preventing spinal cord injury related to the perceptions and behaviors of those involved in the sector. Quality control will be provided by experts in qualitative research and interviews will be stopped when the analyzes will further refine the domains and subdomains. A final framework will be validated to modulate our organization.

ELIGIBILITY:
Inclusion Criteria:

* - Paying patients:
* Spinal cord injured person from any level of injury and any post-traumatic period
* Age 18 to 65 years inclusive
* Person affiliated to the social security or receiving such a plan
* Main ambulation mode: Wheelchair
* Agreeing to participate in interviews

  -- Professional side:
* Medical and paramedical health professionals involved in the care sector or studied various professionals (administrators, insurers, ...) involved in the studied care sector
* Agreeing to participate in interviews

Exclusion Criteria:

* Minors or patients older than 65 years
* Person unable to consent
* Who do not speak the French language
* Person refusing to attend meetings
* Hospitalized person without consent
* Cognitive pathologies incompatible with interviews
* Main wandering mode of patients: walking
* Protected adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of SCI patients recruited in the Physical Medicine and Nantes University Hospital Rehabilitation 15 to 30 patients will be included. Meanwhile, from 10 to 15 professionals involved in the care sector with SCI Nantes University Hospital (mainly caregivers and administrative staff)
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2015-11; Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Validation of a comprehensive conceptual framework reflecting the perceptions and behaviors of patients and professionals involved in the organization of care | Baseline
  specific conceptual framework of preventive organization of the eschar with SCI from domains and subdomains reflecting the perceptions and behaviors of patients and professionals applicable to organizational changes in the medical care of spinal cord injury .

CONTACTS AND LOCATIONS:
Overall Officials: Marc LE FORT, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, Loire Atlantique, France